CLINICAL TRIAL: NCT00126854
Title: High Field (3 Tesla) Magnetic Resonance Spectroscopy Imaging for Follow Up of Prostate Cancer Post Permanent Iodine 125 Brachytherapy Implantation
Brief Title: High Field Magnetic Resonance Spectroscopy Imaging for Follow Up of Prostate Cancer Post Brachytherapy Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA-15-0003 / 22011
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Prostatic Neoplasm
Keywords: brachytherapy; magnetic resonance spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy Imaging

SUMMARY:
The purpose of this study is to establish the correct scanning parameters for obtaining good quality 3 Tesla (3T) magnetic resonance spectroscopy images (MRSI) of the prostate gland before and after brachytherapy implantation for prostate cancer. Three Tesla MRSI may be a valuable additional diagnostic and follow-up investigation for prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for prostate brachytherapy to treat prostate cancer
* Patient signs a study consent form

Exclusion Criteria:

* Have received other radiotherapy for prostate cancer or hormone treatments
* Has contraindication to MRSI scanning
* Does not sign study consent form

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
pilot study meant to establish scanning parameters on 3T MRSI

SECONDARY OUTCOMES:
safety/toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada